CLINICAL TRIAL: NCT06581874
Title: Evaluation of a Collaborative Mental Health Care System
Acronym: MED@PSY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-CHITS-005; 2024-A01115-42 (Other: ID-RCB)
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Psychiatric Adults Patients
Keywords: psychiatry; outpatient follow-up; emergency; ehealth; collaborative care
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emergency (Sham Comparator): Adult patients presenting to the emergency department of the Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer, whether or not referred by their general practitioner.
  Interventions: Other: Clinical assessment by emergency psychiatrist
- Med@Psy Platform (Experimental): Adult patients referred by their general practioner for a psychiatric consultation via the med@psy system.
  Interventions: Other: Psychiatric consultation booked through Med@Psy platform

INTERVENTIONS:
Other: Clinical assessment by emergency psychiatrist — After a clinical assessment by the emergency department psychiatrist which does not lead to hospitalization, the patient will be given a psychiatric interview and sent home.
  Arms: Emergency
Other: Psychiatric consultation booked through Med@Psy platform — The patient will be seen within 48 hours after the consultation with his or her general practitioner by a psychiatrist taking part in the study.
  Arms: Med@Psy Platform

SUMMARY:
In the absence of easy access to second-line ambulatory care, the number of 'inappropriate' psychiatric emergency visits is increasing, with emergency departments becoming the gateway to mental health care.

This is the context in which the 'med@psy' system was set up in the Toulon-Provence-Mediterranean metropolitan area by a private psychiatrist. It facilitates access to psychiatric second referral for General Practitioners (GPs) by pooling the 48-hour supply of psychiatric consultations in real time. It is assumed that this system will facilitate access to outpatient psychiatric care and help to optimize the organisation of patient care and follow-up. The aim of this study is to evaluate the med@psy system in the care pathway for patients with psychiatric disorders.

This study main objective is to compare the proportion of patients with a psychiatric disorder who will receive outpatient follow-up 1 month after a visit to a psychiatric emergency department without hospitalization (Group 1) versus 1 month after a consultation with a psychiatrist within 48 hours via the med@psy system (Group 2).

DETAILED DESCRIPTION:
General practitioners (GPs) are the gateway to the healthcare system and therefore the first point of contact for mental health. A significant proportion of psychiatric disorders can be treated in primary care if GPs have easy access to psychiatric support. However, they are faced with difficulties in accessing secondary care. Around 9/10 consider that it is more difficult to obtain specialist advice than for other disciplines, and say they have difficulty referring a patient for mental health care.

In the absence of easy access to second-line ambulatory care, the number of 'inappropriate' psychiatric emergency visits is increasing, with emergency departments becoming the gateway to mental health care. It is recognized that the deployment of earlier and more graduated care reduces the intensity of disorders, prescriptions for time off work and psychotropic drugs, and hospitalizations.

A new, more preventive, efficient and cost-effective approach to mental health is emerging, with psychiatrists working closely with GPs. This is the context in which the 'med@psy' system was set up in the Toulon-Provence-Mediterranean metropolitan area by a private psychiatrist. It facilitates access to psychiatric second referral for GPs by pooling the 48-hour supply of psychiatric consultations in real time. We assume that this system will facilitate access to outpatient psychiatric care and help to optimize the organisation of patient care and follow-up. The aim of this study is to evaluate the med@psy system in the care pathway for patients with psychiatric disorders.

This study main objective is to compare the proportion of patients with a psychiatric disorder who will received outpatient follow-up 1 month after a visit to a psychiatric emergency department without hospitalization (Group 1) versus 1 month after a consultation with a psychiatrist within 48 hours via the med@psy system (Group 2).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years ;
* Patient presenting to the Centre hospitalier de Toulon La Seyne sur Mer emergency department, with or without referral, and receiving psychiatric advice with discharge without hospitalization after clinical assessment (Group 1) or patients referred for psychiatric consultation via the Med@psy system (Group 2).
* Patient with indication for outpatient follow-up
* Patient with open social security rights

Exclusion Criteria:

* Patient's refusal to take part in research ;
* Patient currently being followed by a psychiatrist. Psychiatric follow-up is defined as at least one consultation with a psychiatrist in the last 3 months, outside an unscheduled care consultation or in an emergency department;
* Patients referred for a suicide attempt, violent or non-violent, serious or non-serious;
* Patients without a declared general practioner;
* Patients already included in the study;
* Patients who do not speak French;
* Patients under judicial protection (guardianship, curatorship, etc.) or safeguard of justice;
* Patient under compulsory care, under a care order or deprived of liberty.
* Any other reason which, in the investigator's opinion, could interfere

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients with a consultation with a psychiatrist, a psychologist or a general practioner one month after the consultation via the med@psy system or the visit to emergency department | 1 month
  Setting up outpatient follow-up from a binary point of view (outpatient follow-up absent or present). This will be defined by whether or not each group has had at least one consultation with a psychiatrist (apart from emergency psychiatric consultations or psychiatric consultations set up at 48 hours with the system), a psychologist or a general practitioner.
  It will be evaluated by means of a telephone survey carried out among patients 1 month after consultation with a psychiatrist via the med@psy system or a visit to the emergency department.

SECONDARY OUTCOMES:
Outpatient follow-up at three months | 3 months
  Outpatient follow-up will be evaluated by the proportion of patients who have had at least one consultation with a psychiatrist, psychologist or general practitioner, in each group, by means of a telephone survey carried out with patients 3 months after the consultation or visit to the emergency department.
Medical partners commitment (part 1) | 1 year
  Medical partners commitment will be assessed by the number of GPs and psychiatrists registered in the Med@psy program.
Medical partners commitment (part 2) | 1 year
  Medical partners commitment will be assessed by the number of patients treated via the program.
Medical partners commitment (part 3) | 1 year
  Medical partners commitment will be assessed by the frequency of use of Med@psy program.
Medical partners commitment (part 4) | 1 year
  Medical partners commitment will be assessed by the average time between referral by the GPs and the psychiatric consultations offered through the Med@psy program, 12 months after its start of use.
Med@psy platform patients characteristics | 1 month
  Description of the patient population who get a psychiatric consultation within 48 hours through the Med@psy platform but who don't come to the consultation. The elements which will be evaluated are : age, sex, place of residence, pathology and reason for referral by a GP.
Functioning Global Assessment | 3 months
  Overall psychological, social and professional functioning will be assessed using the Global Assessment of Functioning (GAF), which will be carried out by a psychologist during a teleconsultation with the patient at 1 and 3 months. Each time, GAF score will be assessed by a second psychologist on the basis of teleconsultation report and the two scores calculated will be compared. In case of different conclusions, the average of the two scores will be taken into account. GAF is a scale used to rate how serious a mental illness may be. It measures how much a person's symptoms affect their day-to-day life on a scale of 0 to 100. 100 corresponds to a better ability to handle daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Korrichi, MD, Study Director
Locations (2):
- France (2):
  - Cabinet médical Korrichi (Med@psy program linked to this office), Toulon, Var
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer emergency reception service, Toulon, Var

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Truelove S, Ng V, Kates N, Alloo J, Sunderji N, Patriquin MJ. Les soins de sante mentale en collaboration: Mobiliser les systemes de sante pour soutenir une approche d'equipe. Can Fam Physician. 2023 Feb;69(2):86-88. doi: 10.46747/cfp.690286. No abstract available. French. PMID 36813512
- [Background] Jones SH, Thornicroft G, Coffey M, Dunn G. A brief mental health outcome scale-reliability and validity of the Global Assessment of Functioning (GAF). Br J Psychiatry. 1995 May;166(5):654-9. doi: 10.1192/bjp.166.5.654. PMID 7620753
- [Background] Kates N, Arroll B, Currie E, Hanlon C, Gask L, Klasen H, Meadows G, Rukundo G, Sunderji N, Ruud T, Williams M. Improving collaboration between primary care and mental health services. World J Biol Psychiatry. 2019 Dec;20(10):748-765. doi: 10.1080/15622975.2018.1471218. Epub 2018 Jun 20. PMID 29722600